CLINICAL TRIAL: NCT04438291
Title: Effects of a Multidisciplinary Team-led School-based Human Papillomavirus Vaccination Health-promotion Programme (MDL-SHPVP) on Improving Vaccine Acceptance and Uptake Among Female Adolescents: A Cluster Randomised Controlled Trial
Brief Title: HPV Vaccination Health-promotion Programme on Vaccine Acceptance and Uptake Among Female Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chau Pak Chun Janita, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14606919
Record Dates: First submitted 2020-06-12; First posted 2020-06-18 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: HPV Infection; Health Behavior; Health Attitude
MeSH Terms: conditions — Papillomavirus Infections; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention schools (Experimental): A 2-hour education session with multicomponent interventions including education sessions with small group dialogues with a registered nurse and trained healthcare and lay volunteers and educational computer games
  Interventions: Other: MDL-SHPVP
- Control schools (Other): Control and usual care
  Interventions: Other: 30-minute educational video

INTERVENTIONS:
Other: MDL-SHPVP — A 2-hour education session with multicomponent interventions including education sessions with small group dialogues with a registered nurse and trained healthcare and lay volunteers and educational computer games
  Arms: Intervention schools
Other: 30-minute educational video — A 30-minute education video (DVD) on HPV, cervical cancer and the HPV vaccine that is designed to enhance HPV vaccine acceptance
  Arms: Control schools

SUMMARY:
The MDL-SHPVP will be developed and a clustered randomised controlled trial will be conducted to evaluate the effects of the MDL-SHPVP and to examine whether the effect of the MDL-SHPVP on the rate of HPV vaccine uptake 1 year after intervention is mediated by parents'/guardians' and female adolescents' HPV knowledge, attitudes and beliefs, adolescents' intention to receive HPV vaccination and vaccine acceptance among their parents/guardians.

DETAILED DESCRIPTION:
2520 adolescents and their parents or guardians from 18 local secondary day schools will be recruited. Multicomponent interventions will be offered to the intervention schools. To build and strengthen the community capacity in health promotion, a team of volunteers will be established to raise awareness of HPV, cervical cancer and HPV vaccine.

Data will be collected at baseline, 1 month and 1 year after intervention. The mixed-effects model will be used to compare the differential changes for each of the primary and secondary outcomes across time between the two groups.

The project is expected to instil a more accurate understanding of HPV and HPV vaccination and support the decision to undergo vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age 14-17 years;

Exclusion Criteria:

* Have received the HPV vaccination before

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The HPV vaccination mainly targets at female in Hong Kong, with the inclusion in Hong Kong Child Immunisation Programme to eligible female students at Primary 5 and 6 from 2019/2020 school year.
Enrollment: 1340 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Female adolescents' uptake of the HPV vaccine | 1 year post-intervention
  Self report uptake of the HPV vaccine by the female adolescents in the past 12 months.

SECONDARY OUTCOMES:
Change of female adolescents' intention to receive HPV vaccination | baseline, 1 month post-intervention
  A 10-point Likert scale will be used to measure the intention indicates "Definitely". 1 indicates "Definitely not" and 10 indicates "Definitely". Higher value means higher intention.
Change of vaccine acceptance among parents/guardians | baseline, 1 month post-intervention
  Precaution Adoption Process Model will be used to measure the vaccine acceptance.
Change of female adolescents' and parents'/ guardians' HPV knowledge | baseline, 1 month post-intervention
  HPV General and HPV Vaccine Knowledge Scale will be used to measure the knowledge.1 point will be given to each correct answer and 0 points will be given to each incorrect or "Don't know" answer. Higher scores mean more HPV knowledge.
Change of female adolescents' HPV attitudes and beliefs | baseline, 1 month post-intervention
  Carolina HPV Immunisation Attitudes and Beliefs Scale will be used to measure the attitudes and belief.
  An 11-point Likert scale will be used, with 0, 5, 7 and 10 indicate "strongly disagree," "somewhat disagree," "somewhat agree" and "strongly agree" respectively, or indicate "extremely ineffective, "somewhat ineffective," "somewhat effective" and "extremely effective" respectively. Higher values mean stronger agreement with the statement and less agreement with or endorsement of HPV vaccination. Five items will be reverse-coded.
Change of parents'/ guardians' HPV attitudes and beliefs | baseline, 1 month post-intervention
  Carolina HPV Immunisation Attitudes and Beliefs Scale will be used to measure the attitudes and belief.
  A 4-point Likert scale will be used. 1,2,3 and 4 indicate "strongly disagree," "somewhat disagree," somewhat agree," and "strongly agree" respectively. Higher values indicate stronger agreement with the statement.

CONTACTS AND LOCATIONS:
Overall Officials: Pak Chun Janita Chau, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo SHS, Chau JPC, Choi KC, Butt L, Lui GCY, Lee VWY, Lau AYL. Effects of an educational health promotion intervention to improve human papillomavirus vaccination acceptance and uptake among adolescent girls: a cluster randomized controlled trial. BMC Public Health. 2025 Oct 9;25(1):3419. doi: 10.1186/s12889-025-24511-4. PMID 41068722
- [Derived] Chau JPC, Lo SHS, Choi KC, Lee VWY, Lui GCY, Chan KM, Lau AYL. Effects of a multidisciplinary team-led school-based human papillomavirus vaccination health-promotion programme on improving vaccine acceptance and uptake among female adolescents: A cluster randomized controlled trial. Medicine (Baltimore). 2020 Sep 11;99(37):e22072. doi: 10.1097/MD.0000000000022072. PMID 32925744